CLINICAL TRIAL: NCT04682431
Title: A Phase 1a/1b Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PY159 as a Single Agent and In Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1a/1b FIH Study of PY159 and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor business decision.
Sponsor: Ikena Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PY159-2-01
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor; Gynecologic Cancer; Breast Cancer; Colorectal Cancer; Gastric Adenocarcinoma; Lung Adenocarcinoma; Pancreatic Cancer; Head and Neck Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Adenocarcinoma of Lung; Pancreatic Neoplasms; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part A: Dose escalation of PY159 alone and in combination with pembrolizumab in a standard 3+3 design; Part B: Dose expansion of one or more dose levels of PY159 administered alone and in combination with pembrolizumab for predefined tumor histology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part A: PY159 Single agent dose level 1 (Experimental): PY159 dose level 1 IV administration, Q3 weekly until consent withdrawal, intolerable toxicity or investigator decision.
  Interventions: Drug: PY159 Single agent dose level 1
- Part A: PY159 Single agent dose level 2 (Experimental): PY159 dose level 2
  Interventions: Drug: PY159 Single agent dose level 2
- Part A: PY159 single agent dose level 3 (Experimental): PY159 dose level 3
  Interventions: Drug: PY159 Single agent dose level 3
- Part A: PY159 single agent dose level 4 (Experimental): PY159 dose level 4
  Interventions: Drug: PY159 Single agent dose level 4
- Part A: PY159 single agent dose level 5 (Experimental): PY159 dose level 5
  Interventions: Drug: PY159 Single agent dose level 5
- Part A: PY159 single agent dose level 6 (Experimental): PY159 dose level 6
  Interventions: Drug: PY159 Single agent dose level 6
- Part A: PY159 single agent dose level 7 (Experimental): PY159 dose level 7
  Interventions: Drug: PY159 Single agent dose level 7
- Part A: PY159/Pembrolizumab Combination dose level 1 (Experimental): PY159 dose level 1 in combination with pembrolizumab
  Interventions: Drug: PY159/Pembrolizumab Combination dose level 1
- Part A: PY159/Pembrolizumab Combination dose level 2 (Experimental): PY159 dose level 2 in combination with pembrolizumab
  Interventions: Drug: PY159/Pembrolizumab Combination dose level 2
- Part A: PY159/Pembrolizumab Combination dose level 3 (Experimental): PY159 dose level 3 in combination with pembrolizumab
  Interventions: Drug: PY159/Pembrolizumab Combination dose level 3
- Part A: PY159/Pembrolizumab Combination dose level 4 (Experimental): PY159 dose level 4 in combination with pembrolizumab
  Interventions: Drug: PY159/Pembrolizumab Combination dose level 4
- PY159 Part B: Single agent dose expansion cohort(s) (Experimental): PY159 Single agent dose expansion cohort(s)
  Interventions: Drug: PY159 Single agent dose expansion cohort
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 1 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 1 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 1
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 2 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 2 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 2
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 3 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 3 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 3
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 4 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 4 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 4
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 5 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 5 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 5
- PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 6 (Experimental): PY159 in combination with pembrolizumab dose expansion cohort 6 to further explore and characterize the anti-tumor activity of PY159 alone and in combination with pembrolizumab in subjects with selected prespecified tumor histologies and known TREM1 expression.
  Interventions: Drug: PY159/Pembrolizumab Combination dose expansion cohort 6

INTERVENTIONS:
Drug: PY159 Single agent dose level 1 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 Single agent dose level 1
Drug: PY159 Single agent dose level 2 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 Single agent dose level 2
Drug: PY159 Single agent dose level 3 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 single agent dose level 3
Drug: PY159 Single agent dose level 4 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 single agent dose level 4
Drug: PY159 Single agent dose level 5 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 single agent dose level 5
Drug: PY159 Single agent dose level 6 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 single agent dose level 6
Drug: PY159 Single agent dose level 7 — Dose of PY159 as a single agent given in a standard 3+3 design.
  Other Names: PY159
  Arms: Part A: PY159 single agent dose level 7
Drug: PY159/Pembrolizumab Combination dose level 1 — Dose of PY159 and given in combination with pembrolizumab
  Other Names: PY159; Pembrolizumab
  Arms: Part A: PY159/Pembrolizumab Combination dose level 1
Drug: PY159/Pembrolizumab Combination dose level 2 — Dose of PY159 and given in combination with pembrolizumab
  Other Names: PY159; Pembrolizumab
  Arms: Part A: PY159/Pembrolizumab Combination dose level 2
Drug: PY159/Pembrolizumab Combination dose level 3 — Dose of PY159 and given in combination with pembrolizumab
  Other Names: PY159; Pembrolizumab
  Arms: Part A: PY159/Pembrolizumab Combination dose level 3
Drug: PY159/Pembrolizumab Combination dose level 4 — Dose of PY159 and given in combination with pembrolizumab
  Other Names: PY159; Pembrolizumab
  Arms: Part A: PY159/Pembrolizumab Combination dose level 4
Drug: PY159 Single agent dose expansion cohort — Dose of PY159 as a single agent given for predefined tumor histology
  Other Names: PY159
  Arms: PY159 Part B: Single agent dose expansion cohort(s)
Drug: PY159/Pembrolizumab Combination dose expansion cohort 1 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 1
Drug: PY159/Pembrolizumab Combination dose expansion cohort 2 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 2
Drug: PY159/Pembrolizumab Combination dose expansion cohort 3 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 3
Drug: PY159/Pembrolizumab Combination dose expansion cohort 4 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 4
Drug: PY159/Pembrolizumab Combination dose expansion cohort 5 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 5
Drug: PY159/Pembrolizumab Combination dose expansion cohort 6 — Dose of PY159 as a single agent and in combination with pembrolizumab for predefined tumor histology
  Other Names: PY159; Pembrolizumab
  Arms: PY159 Part B: PY159/Pembrolizumab Combination dose expansion cohort 6

SUMMARY:
This is an open-label, multicenter, First-In-Human (FIH), Phase 1a/1b study of PY159 in subjects with locally advanced (unresectable) and/or metastatic solid tumors that are refractory or relapsed to Standard Of Care (including Checkpoint Inhibitors, if approved for that indication).

DETAILED DESCRIPTION:
Part A: Dose escalation of PY159 alone and in combination with pembrolizumab in a standard 3+3 design Part B: Dose expansion of one or more dose levels of PY159 administered alone and in combination with pembrolizumab for predefined tumor histology

ELIGIBILITY:
KEY ELIGIBILITY CRITERIA Inclusion Criteria

* Adults ≥18 years of age at the time of study consent
* Subjects with any of the following eligible solid tumor diagnoses as confirmed by cytology or histology. Escalation Cohorts (Part A): Subjects with advanced solid tumors from pre-specified tumor types:

  * head and neck [squamous cell carcinoma, salivary gland, thyroid],
  * gynecologic [including ovarian, fallopian, primary peritoneal, endometrial, cervical, uterine, vaginal, vulvar],
  * pancreatic [adenocarcinoma],
  * lung [adenocarcinoma and squamous cell carcinoma] who are recurrent or refractory to platinum-based chemotherapy in addition to prior treatment with CPI Programmed Cell Death-1 (PD-1)/Programmed Cell Death-Ligand 1 (PD-L1) or who give informed consent to forego such therapy,
  * gastric and esophagogastric junction adenocarcinomas [MSI low and CPI refractory MSI high],
  * breast [TNBC and HR+, HER2-] with metastatic disease that is relapsed or refractory to at least one line of post adjuvant therapy (including a CPI-either alone or in combination, if approved for that indication, and not eligible for other targeted therapies specific for their tumor type).
* Subjects must provide an original, diagnostic tumor sample to determine TREM1 expression (sites have verified source prior to screening and availability of archival tissue during screening). For Part A subjects without an archival tissue sample will only be eligible if they choose and consent to provide a CNB of a primary or metastatic lesion.
* Subjects must have documented radiographic disease progression that include prior treatment with a CPI (alone or in combination), if approved for that indication.
* There is no limit to the number of prior treatments
* Measurable disease by RECIST 1.1.
* All acute toxic effects of any prior antitumor therapy, including immunotherapy, have resolved to Grade < 2 before the start of study drug dosing (except for alopecia or peripheral neuropathy which may be Grade <2 or medication controlled thyroid replacement therapy).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.

Exclusion Criteria

* Subject is a candidate for approved molecularly targeted therapy (e.g., drugs targeting EGFR,VEGF, ALK, ROS-1, NTRK, MET, RET, and BRAF V600E, HER2). Applies to enrolled subjects on both Part A and Part B of the study.
* History of autoimmune disorder requiring ongoing or intermittent disease-modifying therapy excluding thyroid disease well controlled on replacement therapy.
* Untreated and/or uncontrolled brain metastases Stable treated or asymptomatic brain metastases (for at least 1 month prior to enrollment may be enrolled. Subjects with stable treated or asymptomatic brain metastases receiving glucocorticoids must be on a stable dose [≤ 2 mg/day of dexamethasone or an equivalent glucocorticoid] for a minimum of 1month prior to enrollment.)
* Uncontrolled intercurrent illness including, but not limited to, active SARS-CoV-2 infection, active or chronic bleeding event within 28 days prior to first dose of study drug or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician.
* Decompensated liver disease as evidenced by hepatic encephalopathy or coagulopathy.
* Active angina or Class III or IV Congestive Heart Failure (CHF) (NYHA CHF Functional Classification System) or clinically significant cardiac disease within 12 months of first dose. of study drug, including MI, unstable angina, Grade 2 or greater peripheral vascular disease, uncontrolled HTN, or arrhythmias not controlled by medication.
* Any anti-cancer therapy, including small molecules, immunotherapy, chemotherapy, monoclonal antibody therapy (with the exception of bone-modifying agents as supportive care), radiotherapy or any other agents to treat cancer within 14-21 days (dependent upon the agent and drug half-life) of first dose of study drug. Subjects with a prior history of prostate cancer on LHRH agonist are eligible provided they have no evidence of metastatic disease.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | 36 months
  Adverse Events will be summarized by MedDRA system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment related AEs, Serious Adverse Events (SAEs), discontinuations due to AEs, and AEs of at least NCI CTCAE grade 3 severity.
Dose Limiting Toxicity of PY159 (Part A only) | 21 days
  Evaluation of dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Measure PY159 concentration at the end of infusion (CEOI) | 36 months
  Measure PY159 concentration at the end of infusion (CEOI) after the first dose.
Measure PY159 maximum concentration (Cmax) | 36 months
  Measure PY159 maximum concentration (Cmax) at various time points during Cycle 1. All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled pharmacokinetics (PK) time point after start of dosing.
Measure PY159 concentration at the trough level (Ctrough) | 36 months
  Measure PY159 concentration at the trough level (Ctrough). All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled PK time point after start of dosing.
Measure PY159 Area under the curve (AUC)0-t | 36 months
  Measure PY159 Area under the curve (AUC)0-t. All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY159 half-life (T1/2) | 36 months
  Measure PY159 half-life (T1/2). All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY159 Clearance (CL) | 36 months
  Measure PY159 Clearance (CL). All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Measure PY159 Volume at Steady State (Vss) | 36 months
  Measure PY159 Volume at Steady State (Vss). All subjects who received at least 1 dose of PY159 and have at least 1 measured concentration at a scheduled PK time point after start of dosing for at least 1 PK analyte.
Incidence of Anti-Drug Antibody (ADA) formation to PY159 | 36 months
  To evaluate the incidence of anti-drug antibody (ADA) formation to PY159
Determining PY159 time to maximum concentration (Tmax) | 36 months
  Determining PY159 time to maximum concentration (Tmax) during Cycle 1.
Objective response rate (ORR) | 36 months
  The incidents of ORR is defined as either a complete or partial response (PR) per RECIST. Subjects with no baseline data will be considered no responders. ORR will be summarized by dose, tumor type, and overall. ORR will be summarized descriptively.
Clinical Benefit Rate (CBR) | 36 months
  Defined as the percentage of subjects who have achieved complete response (CR), partial response (PR) and stable disease (SD).
Duration of response (DOR) | 36 months
  DOR will be calculated to determine durability. DOR will be measured from the time by which the criteria for CR or PR-whichever is recorded first-are met until the first date by which recurrent or progressive disease is objectively documented. DOR will be assessed using KAPLAN-MEIER methods.

OTHER OUTCOMES:
Progress free survival (PFS) | 36 months
  PFS will be measure from entry onto the study until disease progression or death from any cause. PFS will be assessed using KAPLAN-MEIER methods.
Overall survival (OS) | 36 months
  The duration of overall survival (OS) will be measured from the time of first study drug administration until the date of death. OS will be assessed using KAPLAN-MEIER methods.

CONTACTS AND LOCATIONS:
Overall Officials: Len Reyno, MD, Study Director — Ikena Oncology; Marc Chamberlain, MD, Study Director — Ikena Oncology
Locations (17):
- United States (17):
  - USC Norris Cancer Center, Los Angeles, California
  - UCSF Mount Zion Cancer Center, San Francisco, California
  - UCLA Parkside Cancer Center, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Florida Cancer Specialists - Sarasota - SCRI, Sarasota, Florida
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Case Western Reserve University, Cleveland, Ohio
  - The University of Oklahoma, Norman, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Start South Texas Accelerated Research Therapeutic, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan Y, Xu Y, Huo Z, Zhang H, Peng L, Jiang X, Thomson AW, Dai H. Role of triggering receptor expressed on myeloid cells-1 in kidney diseases: A biomarker and potential therapeutic target. Chin Med J (Engl). 2024 Jul 20;137(14):1663-1673. doi: 10.1097/CM9.0000000000003197. Epub 2024 May 28. PMID 38809056